CLINICAL TRIAL: NCT01076699
Title: A Phase 2, Randomized, Multi-Center, Double-Blind, Placebo-Controlled, Four-Arm Trial to Evaluate the Safety and Efficacy of 3 Different Doses of RVX-100 Versus Placebo for the Treatment of Abdominal Pain in Patients With Irritable Bowel Syndrome Accompanied by Diarrhea (IBS-D)
Brief Title: A Four Arm Study to Evaluate the Safety and Efficacy of 3 Different Doses of RVX-100 Versus Placebo in Subjects With Irritable Bowel Syndrome Accompanied by Diarrhea (IBS-D)
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: recruiting/enrolling participants has halted prematurely but potentially will resume Oct
Sponsor: Revogenex, Inc. (Industry)
Responsible Party: George Kottayil, Chief Operations Officer, Revogenex
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVG-09-005
Record Dates: First submitted 2009-12-01; First posted 2010-02-26 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2010-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: abdominal pain; bloating; diarrhea; irritable bowel
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain; Diarrhea | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group taking 0.075 mg RVX-100 (Active Comparator): This group is taking 0.075 mg RVX-100
  Interventions: Drug: 0.075 mg RVX-100
- Group taking 0.125 mg RVX-100 (Active Comparator): This group is taking 0.125 mg RVX-100
  Interventions: Drug: 0.125 mg RVX-100
- 0.250 mg RVX-100 (Active Comparator): This group is taking 0.250 mg RVX-100
  Interventions: Drug: 0.250 mg RVX-100
- placebo (Placebo Comparator): This group is taking a placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 0.075 mg RVX-100 — This group is taking the lowest dose of RVX-100
  Arms: Group taking 0.075 mg RVX-100
Drug: 0.125 mg RVX-100 — This group is taking an average dose of RVX-100
  Arms: Group taking 0.125 mg RVX-100
Drug: 0.250 mg RVX-100 — This group is taking the highest dose of RVX-100
  Arms: 0.250 mg RVX-100
Drug: placebo — This group is taking a placebo
  Other Names: Sugar pill
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if RVX-100 is safe and effective in treating acute abdominal pain in patients with irritable bowel syndrome accompanied by diarrhea.

ELIGIBILITY:
Inclusion Criteria

* Adult male or female, aged ≥18 and ≤75 years old.
* Subject/ legal representative is able to understand and sign informed consent form.
* Have abdominal pain severity defined as weekly average of "worst abdominal pain in past 24 hours" score of ≥ 3.0 on a 0 to 10 point scale during the second week of the Baseline phase.
* Have IBS-D according to Rome III criteria and ≥25% of stools on the BSS inclusion criteria rated as 6 or 7 during the Baseline phase.
* Not pregnant, lactating, or breastfeeding.
* If a female of childbearing potential, the subject must agree to remain abstinent or practice two medically acceptable forms of contraception during the screening, baseline, treatment, and withdrawal periods. Acceptable forms of contraception include oral contraception, intrauterine devices, implantable devices, and barrier methods. If a barrier method is chosen, a double barrier is required.
* Discontinue all medications used to treat IBS symptoms (prescription and non-prescription) and prescription analgesics at least two (2) weeks prior to the start of the baseline period until after the final study visit. (Final study visit occurs two (2) weeks after the last dose of study medication.) Acetaminophen may be used as a rescue medication as long as it is carefully documented on the Case Report Form (CRF). Fiber supplements are permitted if they are taken at the same frequency and amount throughout the study and were taken during the four (4) weeks prior to the Baseline phase. This must be documented in the source document file and the CRF.
* Willing and able to comply with all study-related procedures, including not incorporating significant changes in diet.

Exclusion Criteria:

* Positive for fecal ova and parasites (O&P) or Clostridium difficile (ELISA) or other bacterial pathogens (standard stool culture) during the Screening phase.
* Taking medication for the treatment of IBS during the baseline phase (other than acetaminophen).
* Taking any treatment for IBS including any of the following classes of medications within 2 weeks prior to baseline visit (Visit 2), or at any point during the study:

  * Antispasmodic or anticholinergic agents
  * Combination products including atropine, hyoscyamine, phenobarbital, and/or scopolamine
  * Antidepressants (such as monoamine oxidase inhibitors [MAOI], selective serotonin reuptake inhibitors [SSRIs], and tricyclic antidepressants), to include, but not limited to the following:
  * Combination products including pheniramine, phenyltoloxamine, or pyrilamine
  * Laxatives
  * Opioids/narcotic analgesics
  * Phenothiazines antipsychotics and anti-emetics
* History of anticholinergic psychosis (psychosis associated with exposure to anticholinergic medications).
* Laboratory values greater than three times the upper limit of normal (ULN) alanine transaminase (ALT/SGPT) or aspartate transaminase (AST/SGOT).
* Laboratory values greater than two times the ULN for total bilirubin (TBil), creatinine (sCr) or blood urea nitrogen (BUN).
* Active infection with hepatitis (A, B, or C) or positive confirmatory test for HIV1, or HIV2 (results of the HIV testing will be kept strictly confidential. Subject may wish to undergo HIV testing as per the guidelines for HIV testing requirements in India pursuant to NACO).
* History of allergic reaction to l-hyoscyamine or atropine, or any component in the formulation of the study drugs.
* Evidence of disease (based on medical history) that could adversely affect the subject's safety during participation in this study or interfere with the interpretation of study results, including but not limited to: glaucoma; pyloric stenosis; clinically significant benign prostatic hypertrophy; clinically significant heart or lung or disease; active peptic ulcer; celiac disease; digestive tract obstruction or paralysis; myasthenia gravis; inflammatory bowel disease; poorly controlled hypertension; hyperthyroidism; decreased hepatic or renal function; urinary retention, or lactose intolerance.
* Use of any investigational drug within 30 days prior to the Baseline Visit (Visit 2), or anytime during study.
* History of non-compliance with treatment or clinical visit attendance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-12 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Change in weekly average abdominal pain severity score from baseline. | 4 weeks

SECONDARY OUTCOMES:
Change in weekly average Abdominal Pain Severity score from baseline to week 8 | 8 weeks
Time to response, based on abdominal pain severity scores. | 8 weeks
Proportion of subjects in each treatment arm who are weekly responders. | 8 weeks
Proportion of subjects in each treatment arm who are end-of-treatment responders | 8 weeks
Number of pain-free days per week, based on responses to the Abdominal Pain Severity scale | 8 weeks
Bowel urgency | 8 weeks
Stool consistency | 8 weeks
Stool frequency | 8 weeks
Fecal incontinence | 8 weeks
Bloating | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hardi, M.D., CPI, Principal Investigator — Metropolitan Gastroenterology Group PC, Chevy Chase Clinical Research
Locations (1):
- Metropolitan Gastroenterology Group, Chevy Chase, Maryland, United States